CLINICAL TRIAL: NCT04496245
Title: Reducing Acute Severe Respiratory Events in Health Care Workers During the Covid-19 Pandemic With OM85
Acronym: COVIDRASP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Griffith University (Other); The Prince Charles Hospital (Other Government); Princess Alexandra Hospital, Brisbane, Australia (Other); Telethon Kids Institute (Other); Queensland Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BV-2020/19
Record Dates: First submitted 2020-07-26; First posted 2020-08-03 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-09

CONDITIONS: Respiratory Viral Infection; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Broncho-Vaxom

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either Group 1 (waitlist control, delayed treatment group) or Group 2 (initial treatment) for treatment for a period of 3 months with 3 months follow-up off treatment
Masking Description: Participants will be randomised to the wait list group (Group 1) or the initial intervention group (Group 2) using a one-to-one ratio, stratified by hospital and department [High risk, lower risk].
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-list control (Active Comparator): One capsule OM85 (7.0 mg) will be given daily for 3 months, commencing in Month 3, with 3 months follow-up off treatment.
  Interventions: Drug: Broncho-Vaxom®
- Initial treatment wtih OM85 (Experimental): One capsule OM85 (7.0 mg) will be given daily for 3 months, commencing on day 0, with 3 months follow-up off treatment.
  Interventions: Drug: Broncho-Vaxom®

INTERVENTIONS:
Drug: Broncho-Vaxom® — Broncho-Vaxom adult capsules® (OM85)
  Other Names: OM85

SUMMARY:
Parallel group, Wait-list design, with treatment delayed for 3 months. Participants will be randomized on a 1:1 ratio with 500 participants per group in Australia.

Group 1: Wait-list control. One capsule OM85 (7.0 mg) will be given daily for 3 months, commencing in Month 3, with 3 months follow-up off treatment.

Group 2: Initial treatment. One capsule OM85 (7.0 mg) will be given daily for 3 months, commencing on day 0, with 3 months follow-up off treatment.

DETAILED DESCRIPTION:
The Covid-19 pandemic has been characterised by acute respiratory distress syndrome (ARDS) accompanied by a systemic cytokine-storm resulting in severe illness, respiratory failure and death in some. Severe Acute Respiratory Syndrome (SARS)- Coronavirus (Cov-2) (COV) infection per se is not the only underlying issue here, as it is becoming evident that ARDS is relatively rare amongst infected subjects, and appears to be associated with gross dysregulation of ensuing host-anti-viral responses resulting in collateral immune-inflammatory-mediated damage to host tissues. Rather than waiting for susceptible subjects to present with COV-associated ARDS, the investigators propose treatment of healthy health care workers (HCW) with a therapeutic agent which simultaneously targets front-line innate anti-viral immune defences, together with the core mechanism that controls immune response intensity in the airways. This research addresses the hypothesis that resistance to development of severe COV-associated respiratory disease in front-line HCW, even in those who develop a primary infection, can be boosted via a regimen of daily dosing with the bacterial-derived immunomodulatory agent OM85.

Aims

1. To demonstrate that daily treatment with OM85 will prevent HCW developing acute respiratory infections (ARI) necessitating removal from the workforce.
2. To elucidate the mechanism of action by which OM85 regulates host immune responses against COV.

Mechanistic studies will primarily test the hypothesis that OM85 pre-treatment modulates the systemic immunoinflammatory response to COV, selectively attenuating potentially pathogenic pro-inflammatory pathways without compromising activation of innate immune pathways central to pathogen clearance. The investigators will additionally collect samples to test the secondary hypothesis that the host response to COV displays uniquely aggressive pro-inflammatory features that differ from those observed with non-COV respiratory infections.

Experimental design: participants will be randomised into two groups; Immediate treatment with OM85 (n=500) or wait-list control with OM85 commencing three months later (n=500). Venous blood samples will be collected from each subject at four time points. Sera will be stored from each time point for assay of COV-specific antibody. For the mechanistic studies the investigators will focus on two groups of subjects who test respectively positive or negative to COV during a defined respiratory illness. These will be further stratified by treatment (OM85 treated (OM+) versus non-treated (OM-) prior to ARI, yielding 4 sets (each n=50) of test samples collected at acute infection which will be utilized for two discrete cross-comparisons: (i) COV+/OM+ versus COV+/OM-, and (ii) COV-/OM+ versus COV-/OM-. Analyses in (i) will be prioritised as they relate exclusively to host-responses to COV and effects of treatment thereon; those in (ii) which will contrast COV-associated response with those elicited by conventional respiratory pathogens and compare respective susceptibility to OM85.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria are eligible for enrolment:

1. HCW in front line clinical departments assessing or caring for patients with suspected or verified COV infection in one of the recruiting hospitals in Brisbane
2. Participants who, in the opinion of the investigator, are able to comply with the protocol for its duration,
3. Written informed consent signed and dated according to local regulations.

Exclusion Criteria:

Participants who meet any of these criteria are not eligible for enrolment:

* Staff with prior COV infection necessitating workforce removal

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Acute Respiratory Infection necessitating workforce removal | 3 months
  The proportion of Health Care Workers contracting an Acute Respiratory Infection necessitating workforce removal in the initial treatment and wait-list control groups assessed at the end of 3 months.

SECONDARY OUTCOMES:
Time to ARI necessitating workforce removal. | 12 months
  The time to the first ARI necessitating workforce removal in the initial treatment and wait-list control groups.
The proportion of Health Care Workers contracting an Acute Respiratory Infection necessitating workforce removal | 12 months
  The proportion of Health Care Workers contracting an Acute Respiratory Infection necessitating workforce removal in the initial treatment and wait-list control groups assessed at the end of 6 and 12 months
The proportion of HCW with documented Cov infection. | 12 months
  The proportion of HCW in the initial treatment and wait-list control group with Cov infection documented by molecular techniques of seroconversion
Time to Lower respiratory infection (LRI) necessitating workforce removal. | 12 months
  The time to the first LRI necessitating workforce removal in the initial treatment and wait-list control groups.
The proportion of Health Care Workers contracting a LRI necessitating workforce removal | 12 months
  The proportion of Health Care Workers contracting LRI necessitating workforce removal in the initial treatment and wait-list control groups assessed at the end of 3, 6 and 12 months
The proportion of HCW with documented Cov LRI. | 12 months
  The proportion of HCW in the initial treatment and wait-list control group with LRI due to Cov infection documented by molecular techniques of seroconversion

CONTACTS AND LOCATIONS:
Overall Officials: PETER D SLY, DSc, Principal Investigator — The University of Queensland
Locations (3):
- Australia (3):
  - The Prince Charles Hospital, Brisbane, Queensland
  - The Princess Alexandra Hospital, Brisbane, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sly PD, Galbraith S, Islam Z, Holt B, Troy N, Holt PG. Primary prevention of severe lower respiratory illnesses in at-risk infants using the immunomodulator OM-85. J Allergy Clin Immunol. 2019 Sep;144(3):870-872.e11. doi: 10.1016/j.jaci.2019.05.032. Epub 2019 Jun 8. No abstract available. PMID 31185221
- [Background] Esposito S, Soto-Martinez ME, Feleszko W, Jones MH, Shen KL, Schaad UB. Nonspecific immunomodulators for recurrent respiratory tract infections, wheezing and asthma in children: a systematic review of mechanistic and clinical evidence. Curr Opin Allergy Clin Immunol. 2018 Jun;18(3):198-209. doi: 10.1097/ACI.0000000000000433. PMID 29561355
- [Background] The Lancet. COVID-19: protecting health-care workers. Lancet. 2020 Mar 21;395(10228):922. doi: 10.1016/S0140-6736(20)30644-9. No abstract available. PMID 32199474

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT04496245/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT04496245/ICF_000.pdf